CLINICAL TRIAL: NCT02339883
Title: Physiological and Psychosomatic Effects of Exposure to MRI Scanning Environment
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150057; 15-N-0057
Record Dates: First submitted 2015-01-15; First posted 2015-01-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-09-27

CONDITIONS: Healthy Volunteers
Keywords: Physiological Measures; MRI; Magnetic Resonance Imaging (MRI); Cognitive Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Magnetic resonance imaging (MRI) creates high-quality images of the human body without x-rays. It uses a strong magnetic field and radio waves to take pictures. Researchers want to test a scanner that uses a high magnetic field strength.

Objective:

- To study how the body responds to being in a high field 11.7T MRI scanner.

Eligibility:

- Healthy people ages 22 65.

Design:

* Participants will be screened with a medical history and physical exam. They will complete a healthy volunteer questionnaire and an MRI safety screening form. They may have a 3T MRI scan of the brain.
* Participants will have an MRI scan. They will lie on a table that will slide in and out of the MRI cylinder very slowly. They will be asked to lie still.
* Participants will do simple tasks while inside the machine. These can include listening and responding to questions, tapping fingers, or moving a hand.
* While in the scanner, participants will hear loud knocking noises. They will get earmuffs.
* Right when they exit the scanner, participants will get a questionnaire to fill out. This will ask about how they felt inside the scanner.
* During the MRI, participants heart rate, respiratory rate, and skin temperature will be measured. Before and after the scan, these things plus blood pressure will be measured.
* Participants will be tested before and after being in the MRI scanner. They will answer questions, take pen-and-paper or computer tests, and do simple actions. Their sense of smell may be tested.

DETAILED DESCRIPTION:
Objective

The goals of this pilot study are to establish a normative database of vital signs, cognitive function and unusual subjective sensations in a 0T scanner. This data will be used as a reference for a future study of the effects of exposure to a 11.7T static magnetic field.

Study Population

26 healthy volunteers, aged 22-65.

Accrual ceiling =50

Accrual Target =26

Drop outs will be replaced

Design

The study consists of one outpatient screening session and one experimental session. Informed consent and a history and neurological examination will be carried out at the screening visit. Vital signs (pulse oximeter, heart rate, respiratory rate and skin temperature) will be measured immediately before and after the experimental scan session, and pulse oximeter, heart rate and respiration will be monitored when the subject is in the scanner. Subjects will remain in the scanner for approximately 1 hour. During the experimental session, while the subject is in the scanner, they will be asked to carry out a brief test of attention at 10-15 minute intervals, up to 3 times during the session. At the end of the experimental session, subjects will fill out the MRI exit questionnaire to rate subjective sensations such as nausea, vertigo, and lightheadedness, on a Likert scale and complete a computerized neuro-cognitive test battery.

Outcome Measures

The objective of the study is to obtain a normative dataset of neuropsychological test measures, physiological parameters, and subjective experiences measures in subjects undergoing 0T exposure.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 22 - 65 years of age
* In good general health
* Able to understand the procedures and requirements and give informed consent
* Fluent in English

EXCLUSION CRITERIA:

All Subjects will answer the NMR safety screening form and the Healthy volunteer form A subject will be excluded if he/she:

* Has any implanted medical device
* Underwent brain surgery, have a central nervous system illness, a neurological lesion or history of neurological or psychiatric disorders
* Medical problems, such as diabetes mellitus, hypertension, pulmonary or airway disease, heart failure, coronary artery disease, history of sleep apnea
* Diagnosable substance dependence
* Consumes more than 1 alcoholic drink per day for women and up to 2 drinks per day for men on a regular basis
* Has any metal in their body due to by trauma or surgery
* Cannot lie comfortably on their back for up to 60 minutes
* Is pregnant
* Have sustained shrapnel injuries
* Has worked as a machinist, or other occupations that have resulted in metal shavings in their eye
* Has claustrophobia
* Has known hearing problems

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12-23; Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Neuropsychological tests | 2 years
Physiological parameters | 2 years
Subjective experience parameters | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Duyn, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)